CLINICAL TRIAL: NCT02968147
Title: High Frequency Jet Ventilation in AF Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PID11559
Record Dates: First submitted 2016-02-01; First posted 2016-11-18 (Estimated); Last update posted 2021-06-01 (Actual); Status verified 2016-11

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; general anaesthesia
MeSH Terms: conditions — Atrial Fibrillation | interventions — High-Frequency Jet Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional ventilation (Experimental): Catheter ablation for persistent atrial fibrillation with general anesthesia and conventional ventilation
  Interventions: Device: Conventional ventilation
- Jet ventilation (Experimental): Catheter ablation for persistent atrial fibrillation with general anesthesia and high frequency jet ventilation
  Interventions: Device: High frequency jet ventilation

INTERVENTIONS:
Device: High frequency jet ventilation — General anaesthesia and ventilation with the Acutronic Monsoon III Jet ventilator system
  Arms: Jet ventilation
Device: Conventional ventilation — General anaesthesia and ventilation with a conventional Phillips intermittent positive pressure ventilator system
  Arms: Conventional ventilation

SUMMARY:
Atrial fibrillation (AF) is a cardiac condition that results in patients experiencing an irregular heart beat resulting in symptoms including palpitations and breathlessness. It is known that in most cases, AF is caused by abnormal electrical activity from the top of the left side of the heart (left atrium) which overrides the heart natural pacemaker in the right atrium. Treatment options include tablets which suppress this abnormal electrical activity, but in some patients these are not sufficient and a procedure is carried out where the areas of abnormal electrical activity are disconnected or 'ablated' to prevent AF from occurring. This treatment is well established and performed worldwide, often under general anaesthetic (GA). The heart and lungs sit close together in the chest, and when the lungs are inflated and deflated during the procedure, the heart also moves. This movement is then transmitted to the special wires or 'catheters' that are placed inside the heart to deliver the ablation treatment. Instability during the treatment can result in ineffective areas of ablation which may later contribute to reduced success of the procedure. Previous research has shown that by reducing the movement of the heart under anaesthesia using alternative techniques can improve catheter stability and improve procedural results. Once such technique is called high frequency jet ventilation (HFJV) which allows the lungs to filled with air using fast and shallow breaths resulting in normal blood oxygen levels with little movement in the heart. This technique has been shown to be safe and effective for this procedure but a direct comparison with conventional ventilation has not been done. The investigators wish to test this and determine if using HFJV improves outcomes during the procedure (i.e. can investigators do the treatment faster and more effectively) and if this translates to better outcomes long term.

DETAILED DESCRIPTION:
Catheter ablation for the treatment of the symptoms of fibrillation is now a well-established technique. The technique is complex and commonly undertaken under general anaesthesia. Catheters are introduced into the circulation from the veins at the top of the leg and advanced to the right side of the heart. Using x-ray and ultrasound guidance, the catheters are passed to the left atrium by puncturing the muscle that divides left and right atria (septum). A model of the left atrium is created and this used to guide the movement of an ablation catheter across the tissue and create ablation lesions that lead to electrical isolation of target sites.

Under general anaesthesia, the lungs are inflated and deflated via the ventilator circuit. The expansion of the lungs results in movement of the heart with each respiratory cycle. This leads to catheter instability as the tissue is moved towards and away from a catheter positioned in the left atrium. This movement is particularly marked at the back of the left atrium. This instability can lead to real time variation in the delivery of energy which can result in ineffective lesions. These will then translate acutely to incomplete isolation and the need for further ablation (thereby increasing procedure time) and later into reconnection of tissue which can result in repeated procedures being needed to achieve an effective outcome. Each procedure carries risk of minor and major complications therefore measures to improve first time success are critical.

Current research supports the use of steerable catheter sheaths (tubes through which the catheters travel to the atria) and 3 dimensional mapping in improving ablation parameters. Data also exists demonstrating significant variation in catheter contact despite these measures. In order to improve catheter stability further, changes to the mode of ventilation has been studied. Small studies have shown that by stopping cardiac movement altogether by transiently stopping ventilation (apnoea) catheter stability is improved and ablation is more effective. However, intermittent apnoea is not an effective method of ventilation in long cases. An alternative is high frequency jet ventilation. This is where the lungs are ventilated with low volume, high speed and high pressure breaths. This technique is well established and has safety data in upper airway surgery and liver radiology procedures where movement of airways and diaphragm needs to be minimized. In view of this, this technique has been studied in AF ablation and has been shown to improve catheter stability and energy delivery with no increase in complications related to the mode of ventilation. However, existing studies have focused mainly in paroxysmal AF patients (where less ablation is needed) and conducted in a non randomized trial design.

The investigators wish to research the use of HFJV in patients undergoing ablation for persistent AF in a prospective and randomised trial to answer the primary and secondary questions shown below.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Indication for left atrial catheter ablation for persistent atrial fibrillation
* Patients may be enrolled in other atrial fibrillation trials at Oxford University Hospitals Foundation Trust (unless directly related to ventilation or ablation strategy)

Exclusion Criteria:

* Age<18 and >85
* Left ventricular ejection fraction <35%
* Severe lung disease - chronic obstructive pulmonary disease or asthma requiring home oxygen therapy or >3 admissions in preceding 12 months
* Previously failed high frequency jet ventilation due to hypercapnia
* Previous catheter ablation for atrial fibrillation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with improved catheter contact force during AF ablation under high frequency jet ventilation | 12 months
  Data will be extracted from the St Jude Medical Velocity/Tacticath system to determine average force (grams/sec) for each applied lesion.

SECONDARY OUTCOMES:
Number of patients with improved lesion power delivery during AF ablation under high frequency jet ventilation | 12 months
  Data will be extracted from the St Jude Medical Velocity/Tacticath system to determine power delivery (force time integral) for each applied lesion.
Number of patients with improved lesion creation during AF ablation under high frequency jet ventilation | 12 months
  Data will be extracted from the St Jude Medical Velocity/Tacticath system to determine power delivery (lesion size index) for each applied lesion.
Number of patients with improved catheter stability during AF ablation under high frequency jet ventilation | 12 months
  Data will be extracted from the St Jude Medical Velocity/Tacticath system to determine catheter movement (mm movement during ablation) for each applied lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Yaver Bashir, MA,DM,FRCP, Study Chair — Clinical Director, Consultant Electrophysiologist
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No